CLINICAL TRIAL: NCT04706130
Title: Rigorous Assessment of P. Vivax Relapses and Primaquine Efficacy for Radical Cure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other); Institut Pasteur du Cambodge (Other)
Responsible Party: Principal Investigator, David Serre, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0010
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Vivax Malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — Primaquine; Artesunate

STUDY DESIGN:
Intervention Model Description: The study will be an open-labelled randomized clinical trial to determine therapeutic efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm1: No primaquine (Other): Enrolled patients will only received blood stage antimalarial (artesunate at 2 mg/kg per day every 24h for 7 days)
  Interventions: Drug: Artesunate
- Arm2: Primaquine low dose (Other): Enrolled patients will received blood stage antimalarial (artesunate at 2 mg/kg per day every 24h for 7 days) and primaquine at 0.25 mg/kg/day for 14 days (starting at day 7)
  Interventions: Drug: Primaquine; Drug: Artesunate
- Arm3: Primaquine high dose (Other): Enrolled patients will received blood stage antimalarial (artesunate at 2 mg/kg per day every 24h for 7 days) and primaquine at 0.50 mg/kg/day for 14 days (starting at day 7)
  Interventions: Drug: Primaquine; Drug: Artesunate

INTERVENTIONS:
Drug: Primaquine — After treatment of the blood stage infection, enrolled participants will receive either no primaquine, a low dose of primaquine or a high dose of primaquine against liver parasites
  Arms: Arm2: Primaquine low dose; Arm3: Primaquine high dose
Drug: Artesunate — All enrolled participants will receive a 7-day treatment of artesunate ((2 mg/kg/day) to clear blood-stage parasites

SUMMARY:
The study will be an open-labelled randomized clinical trial to determine therapeutic efficacy. Note that this will not be an Investigational New Drug application, as only World Health Organization (WHO)-approved drugs will be used at dosage and for conditions approved.

DETAILED DESCRIPTION:
The study will be an open-labelled randomized clinical trial to determine therapeutic efficacy. Note that this will not be an Investigational New Drug application, as only World Health Organization-approved drugs will be used at dosage and for conditions approved.

Eligible patients willing to participate will first be tested prior to enrolment for their glucose-6-phosphate dehydrogenase (G6PD) status by the gold standard spectrophotometric analysis. The investigators will exclude from the study any G6PD deficient (or intermediate females) patient. Treatment allocation will be randomized between i) 7 days of artesunate (2 mg/kg/day for 7 days) alone (Arm1), ii) same artesunate regimen + 0.25 mg/kg/day 14 days of primaquine (Arm2) and iii) same artesunate regimen + 0.5 mg/kg/day 14 days of primaquine (Arm3). All patients will be relocated to a no-transmission city to make sure they are not reinfected during the follow-up. Follow-up will be performed every 24-48h for 90 days. At the end of the follow-up period, all patients that did not receive primaquine (arm1) will be treated according to national guidelines (14 days at 0.25mg/kg/day). Patients will additionally be followed monthly for three months after the end of the relocation.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 and older
* Acute (within 10 days), symptomatic (i.e., history of fever), uncomplicated malaria caused solely by Plasmodium vivax (verified by PCR)
* G6PD normal (as determined by quantitative spectrophotometric assay)

Exclusion Criteria:

* Pregnant, planning to become pregnant or lactating women,
* Received antimalarial drugs in the past month,
* Hb < 8g/dL, < 1,500 neutrophils/μl, or signs of complicated malaria (e.g., vomiting, convulsions,…),
* History of primaquine, artesunate or artesunate-mefloquine allergy or intolerance,
* PCR-positivity for severe acute respiratory syndrome coronavirus 2.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
P. vivax recurrence | 3 months
  Proportion of patients experiencing recurrence as measured by microscopy and PCR and time to recurrence
Markers of P. vivax recurrences | 3 months
  Gene expression or serological markers associated with P. vivax recurrence

SECONDARY OUTCOMES:
Genotypes of relapsing P. vivax parasites | 3 months
  Genotypes of relapsing P. vivax parasites

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Pasteur du Cambodge, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eng V, Lek D, Sin S, Feufack-Donfack LB, Orban A, Salvador J, Seng D, Heng S, Khim N, Tebben K, Flamand C, Sommen C, van der Pluijm RW, White M, Witkowski B, Serre D, Popovici J. 14 days of high-dose versus low-dose primaquine treatment in patients with Plasmodium vivax infection in Cambodia: a randomised, single-centre, open-label efficacy study. Lancet Infect Dis. 2025 Aug;25(8):884-895. doi: 10.1016/S1473-3099(25)00033-7. Epub 2025 Mar 17. PMID 40112852
- [Derived] Eng V, Lek D, Sin S, Feufack-Donfack LB, Orban A, Salvador J, Seng D, Heng S, Khim N, Tebben K, Flamand C, Sommen C, van der Pluijm RW, White M, Witkowski B, Serre D, Popovici J. High versus low dose of 14 days treatment of primaquine in Plasmodium vivax infected patients in Cambodia: a randomised open-label efficacy study. medRxiv [Preprint]. 2025 Jan 2:2025.01.01.25319862. doi: 10.1101/2025.01.01.25319862. PMID 39802788